CLINICAL TRIAL: NCT01034774
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability, Plasma Pharmacokinetics and Lung Penetration of Intravenous (IV) ACHN-490 in Healthy Subjects
Brief Title: Phase 1 Study to Determine Safety, Blood PK and Lung Penetration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACHN-490-003
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Volunteers
Keywords: Human volunteers
MeSH Terms: interventions — plazomicin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACHN-490 Injection (Active Comparator): ACHN-490 Injection will be given either 1 or 5 consecutive days at a dose of 15mg/kg.
  Interventions: Drug: ACHN-490 Injection
- Placebo is Normal Saline (Placebo Comparator): Placebo will be given either 1 or 5 consecutive days to mask when ACHN-490 Injection is given.
  Interventions: Drug: Placebo (normal saline)

INTERVENTIONS:
Drug: ACHN-490 Injection — ACHN-490 Injection at 15mg/kg is given either 1 or 5 consecutive days. Cohort 1 receives 5 consecutive days of treatment and Cohort 2 receives a single dose of treatment.
  Arms: ACHN-490 Injection
Drug: Placebo (normal saline) — Placebo is given at the same volume as ACHN-490 Injection to maintain the blind.
  Other Names: Normal Saline; NS
  Arms: Placebo is Normal Saline

SUMMARY:
Multiple center, double-blind, randomized, placebo-controlled study to see if it is safe to give ACHN-490 Injection for 5 consecutive days, to measure plasma pharmacokinetics, and to determine lung penetration of ACHN-490 (measured in ELF-epithelial lining fluid)after a single dose of ACHN-490 Injection in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women
* Within normal weight limits
* In good health with normal routine laboratory results
* Willing to not use media players (such as MP3 players) or devices with ear pieces and avoid exposure to loud noises

Exclusion Criteria:

* No ongoing medical conditions such as heart disease, high blood pressure, asthma, diabetes, seizures, or kidney problems
* No problems with hearing or balance
* No previous injury or surgery to the ears
* No family history of hearing loss before the age of 65
* Not taking any medications other than birth control medication
* Smokers or use of tobacco products
* Recent blood donors
* No excessive alcohol intake or illegal substances
* No allergy to aminoglycosides (a type of antibiotic)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety measured by reported adverse events after administering ACHN-490 Injection/placebo for 5 consecutive days | Throughout the study

SECONDARY OUTCOMES:
Lung penetration as estimated from ACHN-490 measured in ELF | 1 Day
Plasma pharmacokinetic profile as measured by the concentration of ACHN-490 in the blood after 5 days of dosing | Through 24 hours after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Havrilla, MS, RN, Study Director — Achaogen, Inc.